CLINICAL TRIAL: NCT04687202
Title: The Clinical Characteristics, Management and Prognosis of Patients Developing Intraoperative Cardiac Arrest During Transcatheter Aortic Valve Implantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 研2019-125
Record Dates: First submitted 2020-12-24; First posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Cardiac Arrest, Transcatheter Aortic Valve Implantation
MeSH Terms: conditions — Heart Arrest | interventions — Records

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients developing CA: Including patients developing intraoperative cardiac arrest during transcatheter aortic valve implantation from January 2014 to May 2019
  Interventions: Other: follow up and record

INTERVENTIONS:
Other: follow up and record — None additional intervention was applied to the subjects.

SUMMARY:
This study was aimed to investigate the clinical characteristics, management and prognosis of patients developing intraoperative cardiac arrest during transcatheter aortic valve implantation

ELIGIBILITY:
Inclusion Criteria: patients who developed intraoperative cardiac arrest during transcatheter aortic valve implantation from January 2014 to May 2019 -

Exclusion Criteria: None.

-

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients who developed intraoperative cardiac arrest during transcatheter aortic valve implantation from January 2014 to May 2019
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1month
  In-hospital mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No